CLINICAL TRIAL: NCT03768388
Title: A Phase I Randomized, Open-Label, Two-Period, Two-Sequence Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of Levoketoconazole in Healthy Subjects
Brief Title: Levoketoconazole Food Effect Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortendo AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: COR-2017-02
Record Dates: First submitted 2018-11-30; First posted 2018-12-07 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasting State (Other): A single 600 mg dose of levoketoconazole administered in a fasting state.
  Interventions: Drug: levoketoconazole
- Fed State (Other): A single 600 mg dose of levoketoconazole administered in a fed state.
  Interventions: Drug: levoketoconazole

INTERVENTIONS:
Drug: levoketoconazole — food effect
  Other Names: COR-003

SUMMARY:
This is a phase I, randomized, open-label, single-dose, two-period, two-sequence crossover study in healthy male and female subjects to evaluate the effect of food on the PK of levoketoconazole.

DETAILED DESCRIPTION:
In each period of the randomized, two period crossover study, levoketoconazole will be administered orally as a single dose of 600 mg levoketoconazole to subjects in the fasted state or fed (at 30 minutes after beginning consumption of a standardized high-fat meal). Subjects assigned to one treatment in Period 1 will be assigned to the opposite treatment in Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18-55 years of age, inclusive, at time of consent.
2. Subject has a body mass index (BMI) between 18 and 32 kg/m2, inclusive.
3. Subject is in good general physical health as determined by absence of clinically significant medical history, physical examination findings, vital signs, clinical laboratory evaluations, and ECG measurements.
4. Subject has not consumed and agrees to abstain from taking any prescription drugs, dietary supplements including vitamins and herbal preparations, or non-prescription drugs (except as authorized by the Investigator AND Medical Monitor) for 14 days prior to CRU admission, during washout period, and through Follow-Up.
5. Subject has not consumed alcohol-containing beverages for 3 days prior to CRU admission and agrees not to consume alcohol through Follow-Up.
6. Subject is a nonsmoker (for at least 3 months) with negative urinary cotinine test at Screening and agrees to abstain from tobacco- and nicotine-containing products for the duration of the study.

Exclusion Criteria:

1. Evidence of any out-of-normal-range laboratory value at Screening that has not been reviewed, approved, and documented as Not Clinically Significant by the Investigator.
2. Concurrent medical illness that would interfere with the conduct of the study in the opinion of the Investigator.
3. History or presence of clinically significant cardiovascular, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, psychiatric, renal, hepatic, chronic respiratory, or gastrointestinal disease as judged by the Investigator.
4. Positive urine drug screen for drugs-of-abuse, including cocaine, tetrahydrocannabinol, opioids, benzodiazepines, amphetamines, and barbiturates, and/or positive urine screen for alcohol at Screening and CRU admission.
5. Treatment with an investigational drug within the longer of 30 days or five half-lives of the investigational drug preceding the first dose of study drug.
6. Subject is positive for Human Immunodeficiency Virus (HIV), hepatitis B, and/or hepatitis C on Screening assessments.
7. Subject has an acute illness within 7 days of CRU admission.
8. Subject has donated plasma within 7 days of drug administration.
9. Subject has donated 1 or more pints of blood (or equivalent blood loss) within 30 days prior to drug administration.
10. History of caffeine consumption exceeding 8 cups of coffee/day (1 cup = 8 fluid ounces) within 14 days prior to first dose, or consumption of any caffeine- or chocolate-containing products for 3 days prior to CRU admission each week. Caffeine-containing foods and/or beverages (e.g., tea and cola) should be considered equivalent to coffee.
11. Female subjects who are pregnant or lactating.
12. Males with hemoglobin less than 12.0 g/dL; Females with hemoglobin less than 11.0 g/dL.
13. Subjects who have had difficulties with swallowing whole tablets.
14. Subjects with body habitus preventing repeated venipuncture as required by protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of levoketoconazole | 24 hours
  Maximum observed plasma concentration (Cmax) of levoketoconazole for fed vs. fasted condition
Time to maximum concentration (Tmax) of levoketoconazole | 24 hours
  Time to maximum concentration (Tmax) of levoketoconazole for fed vs. fasted condition
Apparent Terminal Elimination Phase Rate Constant (λz) of levoketoconazole | 24 hours
  Apparent Terminal Elimination Phase Rate Constant (λz) of levoketoconazole for fed vs. fasted condition
Terminal phase half-life (t 1/2) of levoketoconazole | 24 hours
  Terminal phase half-life (t 1/2) of levoketoconazole for fed vs. fasted condition
Area under the plasma concentration-time curve (AUC) of levoketoconazole | 24 hours
  Area under the plasma concentration-time curve (AUC) from time 0 to time of last measurable plasma concentration (AUClast) and from time 0 extrapolated to infinity (AUCinf) of levoketoconazole for fed vs. fasted condition

SECONDARY OUTCOMES:
Incidence of Adverse Events | 14 days
  AEs leading to discontinuation, AEs of Special Interest (AESIs), AEs related to study drug and AE severity will be summarized by study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schoenfeld, MD, Study Director — Cortendo AB
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No